CLINICAL TRIAL: NCT04931459
Title: A Phase 1 Placebo-Controlled, Single- and Multiple-Dose Study of the Safety, Tolerability, and Pharmacokinetics of Intravenous ACU193 in Mild Cognitive Impairment or Mild Dementia Due to Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Blood Levels of ACU193 in Participants With MCI or Mild AD
Acronym: INTERCEPT-AD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acumen Pharmaceuticals (Industry)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACU-001; 3U01AG053247 (NIH)
Record Dates: First submitted 2021-05-18; First posted 2021-06-18 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Diseases; Mild Cognitive Impairment; Mild dementia
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Study ACU-001 is a placebo-controlled study to investigate the safety, tolerability, pharmacokinetics, and pharmacodynamics of single and multiple escalating doses of intravenous ACU193. A two-part single-ascending dose (SAD)/multiple-ascending dose (MAD) study design will be conducted in a population of individuals with early AD (MCI or mild dementia due to AD).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACU193 Administration (Experimental): Participants will receive 1 to 3 doses of ACU193 by intravenous (IV) infusion.
  Interventions: Drug: ACU193
- Placebo Administration (Placebo Comparator): Participants receive 1 to 3 doses of matching ACU193 placebo by intravenous (IV) infusion.
  2 participants per cohort will receive placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACU193 — Intravenous ACU193
  Arms: ACU193 Administration
Drug: Placebo — Intravenous Placebo
  Arms: Placebo Administration

SUMMARY:
This Phase 1 study is a single ascending dose (SAD) and multiple ascending dose (MAD), placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of intravenous ACU193 when administered to participants diagnosed with Mild Cognitive Impairment (MCI) or Mild Dementia due to Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ages 55 to 90 (inclusive).
2. Participant weighs at least 41 kg (90 lbs) and no more than 113 kg (250 lbs) before study drug administration.
3. Female participants must be surgically sterile or be at least two years post-menopausal or at least one year post-menopausal with an elevated follicle stimulating hormone (FSH). Male participants with a female partner of child-bearing potential must use adequate contraception.
4. Individual (or the participant's Legally Authorized Representative [LAR]) is able to give informed consent.
5. Are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
6. Must meet all of the following clinical criteria for MCI due to AD or mild AD at Screening:

   1. Participant meets NIA-Alzheimer's Association (NIA-AA) criteria for MCI due to AD or probable AD.
   2. A global Clinical Dementia Rating (CDR) of 0.5 or 1.0.
   3. A Mini-Mental State Examination (MMSE) score between 18 and 30 (inclusive).
   4. A positive amyloid positron emission tomography (PET) scan.
7. Must consent to apolipoprotein E (APOE) genotyping.
8. If using cholinesterase inhibitors or memantine to treat symptoms related to AD, doses must be stable for at least four weeks prior to Baseline and the participant must be willing to keep the doses stable throughout the duration of the study.
9. Must have a reliable informant or caregiver who is willing and able to perform all caregiver roles as specified in the caregiver Informed Consent Form (ICF).

Exclusion Criteria:

1. Receipt of any investigational biological drug within less than one year of Baseline or of any investigational small molecule drug within less than six months of Baseline. Receipt of any approved treatments that target amyloid plaques in the brain within less than one year of Baseline.
2. Currently receiving or likely to require the following types of anticoagulants: coumarins and indandiones, Factor Xa inhibitors, heparins, thrombin inhibitors.
3. Has known humanized monoclonal antibody allergy or hypersensitivity.
4. History of significant neurological disease, other than AD, that may affect cognition or ability to complete the study, including but not limited to, other dementias, serious infection of the brain, Parkinson´s disease, or adult epilepsy.
5. Has had magnetic resonance imaging (MRI) or computerized tomography (CT) of brain within previous two years showing pathology that would be inconsistent with a diagnosis of AD.
6. Has MRI with results showing greater than four amyloid-related imaging abnormalities hemorrhage/hemosiderin deposition (ARIA-H), presence of any amyloid-related imaging abnormalities edema/effusions (ARIA-E), or superficial siderosis.
7. Has any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or a cardiac pacemaker that is not compatible with MRI.
8. Current serious or unstable clinically important illness that, in the judgment of the Investigator, is likely to affect cognitive assessment including visual and hearing impairment, deteriorate, or affect the participant's safety or ability to complete the study, including psychiatric, hepatic, renal, gastroenterological, respiratory, cardiovascular, endocrinological, immunologic, or hematologic disorders.
9. Has an ongoing or new clinically significant laboratory abnormality, as determined by the Investigator.
10. Has a history or presence of clinically significant abnormal 12-lead electrocardiogram (ECG) or an ECG with QT interval corrected using Fridericia's formula (QTcF) >470 msec for female participants or >450 msec for male participants. As the ECGs are obtained in triplicate and are meant to be interpreted together, if one of the three ECGs in the triplicate has a QTcF above the threshold, eligibility of the participant should be determined based on clinical judgment of the Investigator in consultation with the medical monitor. If two of the three ECGs in the triplicate have a QTcF above the threshold, then the participant would not be eligible.
11. Within one year before Screening, any of the following: myocardial infarction; moderate or severe congestive heart failure, New York Heart Association class III or IV; hospitalization for, or symptom of, unstable angina; syncope due to orthostatic hypotension or unexplained syncope; known significant structural heart disease (eg, significant valvular disease, hypertrophic cardiomyopathy), or hospitalization for arrhythmia.
12. History of seizure, transient ischemic attack (TIA), or stroke within the last 18 months.
13. History of clinically significant carotid or vertebrobasilar stenosis or plaque.
14. History of a malignant disease with the exception of resected cutaneous squamous cell carcinoma in situ, basal cell carcinoma, cervical carcinoma in situ, or in situ prostate cancer with a normal prostate-specific antigen posttreatment within the last five years.
15. Current symptoms meeting Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition, criteria for major depressive disorder or any current primary psychiatric diagnosis other than AD if, in the judgment of the Investigator, the psychiatric disorder or symptom is likely to confound interpretation of drug effect, affect cognitive assessments, or affect the participant´s ability to complete the study.
16. Are a suicide risk, as determined by meeting any of the following criteria:

    1. Suicide attempt within the six months prior to Baseline.
    2. Suicidal ideation as defined by a positive response to Question 5 on the Columbia-Suicide Severity Rating Scale (C-SSRS) suicidal ideation section.
    3. Significant risk of suicide, as judged by the site Investigator.
17. History of multiple concussions, significant head trauma, or objective change in neuropsychological function within the last five years.
18. History of human immunodeficiency virus (HIV).
19. History of alcohol or drug abuse/dependence within the last five years.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence and Nature of Treatment-Related Adverse Events (AE) or Serious Adverse Events (SAE) as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) | Baseline up to 20 weeks (SAD); 14, 18 or 28 weeks (MAD)
  Proportion of participants with AE, discontinuations due to AE or SAE, and withdrawals from the study due to AE
Change in Clinical Laboratory Tests | Baseline up to 20 weeks (SAD); 14, 18 or 28 weeks (MAD)
  Incidence and clinically significant abnormal changes in clinical laboratory assessments (hematology, clinical chemistry, urinalysis)
Changes in 12-Lead ECGs | Baseline up to 20 weeks (SAD); 14, 18 or 28 weeks (MAD)
  Clinically significant abnormal changes in 12-Lead ECGs for PR, QRS, QT, QTcF, and QTcB
Changes in the Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to 20 weeks (SAD); 14, 18 or 28 weeks (MAD)
  Presence of suicidal ideation as defined by a positive response to Question 5 on the C-SSRS suicide ideation section
Changes in Magnetic Resonance Imaging (MRI) | Baseline (predose) up to 20 weeks (SAD); 14, 18 or 28 weeks (MAD)
  Brain magnetic resonance imaging (MRI) findings to assess amyloid-related imaging abnormalities (ARIA), including incidence of ARIA-E (edema) or ARIA-H (hemosiderosis)

SECONDARY OUTCOMES:
Estimate Blood Levels of ACU193 | Up to 140 days post dose
  Area under the concentration-time curve (AUC) from time zero to the time of last measurable concentration (AUCt)
Estimate Maximum Blood Levels of ACU193 | Up to 140 days post dose.
  Maximum observed blood concentration Cmax(obs).
Estimate Time to Reach Maximum Blood Levels of ACU193 | Up to 140 days post dose.
  Time to reach Tmax(obs)
Estimate Blood Levels of ACU193 | Up to 140 days post dose.
  Area under the plasma concentration-time curve from time 0 to infinity (AUC∞)
Estimate Clearance of ACU193 | Up to 140 days post dose
  Clearance (CL)
Estimate Volume of Distribution of ACU193 | Up to 140 days post dose
  Apparent volume of distribution at terminal phase (Vz)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Siemers, MD, Principal Investigator — Acumen Pharmaceuticals, Inc.; Russell Barton, Study Director — Acumen Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Clinical Endpoints, Scottsdale, Arizona
  - Orange County Research Institute, Anaheim, California
  - Hoag Hospital Newport Beach, Newport Beach, California
  - Velocity Clinical Research, Hallandale, Florida
  - Charter Research, Lady Lake, Florida
  - Columbus Clinical Services, Miami, Florida
  - Combined Research Orlando Phase I-IV, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Santos Research Center, Tampa, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, Decatur, Georgia
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Columbia University, New York, New York
  - AMC Research, Matthews, North Carolina
  - Abington Neurological Associates, Abington, Pennsylvania
  - Kerwin Medical Center, Dallas, Texas
  - Clinical Trials Network, Houston, Texas

IPD SHARING:
Plan to Share IPD: No